CLINICAL TRIAL: NCT00393055
Title: Xylitol Adult Caries Trial (X-ACT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Jim Bader, DDS, Res Prof, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NIDCR-18038; U01DE018038 (NIH)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Xylitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- xylitol lozenge (Experimental): 1g xylitol lozenge. Five/day, dissolved in mouth
  Interventions: Dietary Supplement: xylitol
- inactive lozenge (Placebo Comparator): 1g placebo lozenge. Five/day, dissolved in mouth
  Interventions: Dietary Supplement: inactive lozenge

INTERVENTIONS:
Dietary Supplement: xylitol — 1g xylitol lozenges to be dissolved in mouth. Five lozenges daily for three years
  Arms: xylitol lozenge
Dietary Supplement: inactive lozenge — 1g inactive lozenge, dissolved in mouth. Five/day for three years
  Other Names: placebo
  Arms: inactive lozenge

SUMMARY:
The purpose of the trial is to determine the extent to which daily use of xylitol lozenges reduces the appearance of new caries lesions in adults who tend to experience such lesions (i.e., caries-active adults).

DETAILED DESCRIPTION:
Dental caries incidence is higher in adults than children. Recent recommendations from both the Centers for Disease Control and an NIH Consensus Development Conference on dental caries call for clinical trials of caries prevention methods in caries-active adults. Little is known about the effectiveness of caries prevention methods in adults, and virtually no information exists with respect to prevention among adults who are at elevated risk for developing caries lesions. This application describes a clinical trial of an intervention to prevent dental caries in caries-active adults that is responsive to the CDC and Consensus Conference recommendations.

The Xylitol for Adult Caries Trial (X-ACT) is a three-year, multi-center, randomized, placebo-controlled, double-blind study to determine the effectiveness of xylitol lozenges in reducing the incidence of coronal and root caries in caries-active adults. The intervention is the daily use of xylitol lozenges. Participants will be 750 adults (ages 25-75) with current or recent caries lesions who are dental school patients at one of three Clinical Centers in Chapel Hill, NC, Birmingham, AL, and San Antonio TX. These Clinical Centers offer diverse populations with substantial proportions of minority populations that enhance the generalizability of the findings. The Study Chair is located at the University of North Carolina-Chapel Hill, and the Data Coordinating Center is at the Kaiser Permanente Center for Health Research in Portland, OR.

This intervention is being tested because it represents a potentially effective caries prevention method with a high likelihood of adoption by dental practitioners as an "add on" caries preventive method for their caries-active patients. The potential for adoption of the intervention is an important consideration because current data suggest that caries-active adults are underexposed to caries-preventive treatment in dental practices. If effective, the intervention also holds potential as a public health measure.

ELIGIBILITY:
Inclusion Criteria:

* age 25-80
* at least one caries lesion in year prior to enrollment
* at least 12 teeth without crowns
* no allergies to xylitol or aspartame
* anticipate remaining in area for 3 years

Exclusion Criteria:

* 10 or more caries lesions in year prior to enrollment
* currently receiving long-term antibiotic therapy
* history of head and neck radiation

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
combined root and coronal D2FS (dental caries) increment | 3 year

SECONDARY OUTCOMES:
combined root and coronal D12FS (dental caries) increment | three year
separate root and coronal D12FS (dental caries) increments | 3 years
association of lozenge use with D12FS (dental caries) in control group only | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: James D Bader, DDS MPH, Principal Investigator — UNC School of Dentistry
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of North Carolina School of Dentistry, Chapel Hill, North Carolina
  - University of Texas Health Science Center, San Antonio, Texas

REFERENCES:
- [Derived] Brown JP, Amaechi BT, Bader JD, Gilbert GH, Makhija SK, Lozano-Pineda J, Leo MC, Chen C, Vollmer WM; X-ACT Trial Collaborative Group. Visual scoring of non cavitated caries lesions and clinical trial efficiency, testing xylitol in caries-active adults. Community Dent Oral Epidemiol. 2014 Jun;42(3):271-8. doi: 10.1111/cdoe.12082. Epub 2013 Nov 8. PMID 24205951
- [Derived] Ritter AV, Bader JD, Leo MC, Preisser JS, Shugars DA, Vollmer WM, Amaechi BT, Holland JC. Tooth-surface-specific effects of xylitol: randomized trial results. J Dent Res. 2013 Jun;92(6):512-7. doi: 10.1177/0022034513487211. Epub 2013 Apr 15. PMID 23589387
- [Derived] Bader JD, Vollmer WM, Shugars DA, Gilbert GH, Amaechi BT, Brown JP, Laws RL, Funkhouser KA, Makhija SK, Ritter AV, Leo MC. Results from the Xylitol for Adult Caries Trial (X-ACT). J Am Dent Assoc. 2013 Jan;144(1):21-30. doi: 10.14219/jada.archive.2013.0010. PMID 23283923
- [Derived] Bader JD, Shugars DA, Vollmer WM, Gullion CM, Gilbert GH, Amaechi BT, Brown JP. Design of the xylitol for adult caries trial (X-ACT). BMC Oral Health. 2010 Sep 29;10:22. doi: 10.1186/1472-6831-10-22. PMID 20920261